CLINICAL TRIAL: NCT03763487
Title: Marginal Zone Similar to B Lymphocytes in Peripheral Blood in Patients With Celiac Disease
Brief Title: The Aim of This Project is to Verify Whether a Depletion of B Cell Memory Subpopulation ("Marginal-zone-like") CD19 + IgD + CD27 + and CD19 + IgM + CD27 + is a Useful Indicator of Hyposplenism in Patients With Celiac Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Proff. Jan Bures, MD, Principal Investigator, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Indicators of celiac activity
Record Dates: First submitted 2018-10-12; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Celiac Disease
Keywords: celiac sprue, celiac, hyposplenism, IgM memory, B lymphocytes
MeSH Terms: conditions — Celiac Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 50 patients and 30 healthy blood donor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Ultrasound examination: scaled to spleen size (spleen volumetry) Methodology of laboratory tests: venous blood sampling
  Interventions: Diagnostic Test: venous blood sampling; Procedure: spleen volumetry
- healthy blood donors (No Intervention): No intervention in this group.

INTERVENTIONS:
Diagnostic Test: venous blood sampling — Venous blood samples to determine memory B lymphocytes.
  Arms: Patients
Procedure: spleen volumetry — Ultrasound examination of spleen to scaled the size.
  Arms: Patients

SUMMARY:
This project is expected to confirm the hypothesis that hyposplenism in patients with celiac disease is not conditioned by a selective memory deficiency of B lymphocytes.

Other objectives of project are:

* determination of gliadin 33-mer in faecal and urine as indicators patient´s adherence to gluten-free diet
* determination of citrulline in plasma as an indicator of the overall functional capacity enterocytes

DETAILED DESCRIPTION:
Ultrasound examination is focused to spleen size (spleen volumetry). Methodology of laboratory examinations is based on venous blood sampling for the determination of memory B-like marginal zone by flow cytometry; gliadin 33-mer (ELISA) determination in faecal and urine sample; blood plasma extraction for citrulline (high performance liquid chromatography, HPLC).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed celiac disease
* age over 18 years

Exclusion Criteria:

* haematological diseases and cancer
* infectious and non-infectious inflammation of the small intestine
* congenital or acquired immunodeficiency
* autoimmune disease
* immunosuppressant treatment
* diabetes mellitus
* pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
concentration of B-lymphocytes as parameter to evaluate treatment effect | one year
  assessment method: blood sampling, units: the measurement results are in absolute numbers, method: flow cytometry
concentration of B-lymphocytes as parameter to evaluate treatment effect | one year
  assessment method: blood sampling, units: the measurement results are in percentage numbers, method: flow cytometry
concentration of citrullin in plasma as parameter to evaluate treatment effect | one year
  assessment method: blood sampling, units: μmol/l (micromol/l; Citrullin cut-off for intestinal failure is <20μmol / L), method: mass spectrometry (LC-MS instrumentation with internal isotopically labeled standard)
concentration of ornithin in plasma as parameter to evaluate treatment effect | one year
  assessment method: blood sampling, units: μmol/l (micromol/l), method: mass spectrometry (LC-MS instrumentation with internal isotopically labeled standard)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Králové, Hradec Králové, The Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC1419299/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/18270242
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5415212/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/11113071